CLINICAL TRIAL: NCT03240172
Title: Assessment of DNA Damage and Capacity of DNA Repair System Among Nuclear Medicine and Clinical Oncology Workers Exposing to Ionizing Radiation
Brief Title: Assessment of DNA Damage Due to Ionizing Radiation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, asmaa mohamed, Director, clinical research, Assiut University
Other Study IDs: 17200101
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Occupational Exposure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
detection of DNA damage due to occupational exposure to low dose ionizing radiation using comet assay technique and genotyping of certain DNA repair genes to detect inherited polymorphism.

ELIGIBILITY:
Inclusion Criteria:

* • The radiation exposed workers will include nurses, technicians and physicians.

These persons will be occupationally exposed to different radiation sources.

Exclusion Criteria:

* History of diagnostic X-rays, radiotherapy and/or chemotherapy 12 months prior to sampling.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Case control study that will include 100 participants (50 radiation exposed workers will be compared with 50 healthy age and sex-matched control group not exposed to radiation.
  G power program was used to calculate the sample size for two independent groups. power calculation estimated to detect an effect size of 0.88 of difference between means of two independent groups, with a p value < 0.05 and 80% power,.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07-20 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
detection of DNA damage due to occupational exposure to ionizing radiation | 6 month
  comet assay technique will be used

CONTACTS AND LOCATIONS:
Overall Officials: asmaa HA mohamed, PHD, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt